CLINICAL TRIAL: NCT02912676
Title: A Phase 1-2 Study of 6-Thioguanine in Combination With Methotrexate and 6-Mercaptopurine During Maintenance Therapy of Childhood, Adolescent, and Adult Lymphoblastic Non-Hodgkin's Lymphoma and Acute Lymphoblastic Leukemia
Brief Title: Thiopurine EnhAnced Maintenance Therapy
Acronym: TEAM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kjeld Schmiegelow (Other)
Collaborators: Danish Child Cancer Foundation (Other); Nordic Society for Pediatric Hematology and Oncology (Other)
Responsible Party: Sponsor-Investigator, Kjeld Schmiegelow, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rigshospitalet - TEAM
Record Dates: First submitted 2016-09-12; First posted 2016-09-23 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma
Keywords: Cancer; Thioguanine; Acute Lymphoblastic Leukemia; 6 Mercaptopurine; Maintenance Therapy of Leukemia; Denmark; Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms | interventions — Thioguanine; Mercaptopurine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 6TG/6MP/MTX (Experimental): Single arm feasibility study aiming to demonstrate the applicability of combining incremental doses of oral 6-Thioguanine with oral daily 6-Mercaptopurine and oral weekly Methotrexate in order to achieve mean levels of DNA-TG above 500 fmol/mikrogram DNA.
  Interventions: Drug: Thioguanine (oral)

INTERVENTIONS:
Drug: Thioguanine (oral) — Addition of incremental doses of oral Thioguanine to oral daily 6-mercaptopurine and oral weekly methotrexate maintenance therapy of Acute Lymphoblastic Leukemia and Lymphoblastic Lymphoma. Oral 6-thioguanine is added at a starting dose of 2.5 mg/m.sq. with dose increments of 2.5 mg/m.sq. at two weeks intervals until a maximum dose of 12.5 mg/m.sq. of 6-thioguanine is given or dose-limiting toxicity occurs.
  Other Names: 6-mercaptopurine (oral); Methotrexate (oral)

SUMMARY:
Acute Lymphoblastic Leukaemia (ALL) is the most frequent cancer in children. The survival rate has improved significantly during the last decades, but the treatment still fails to cure 15 % of the patients. Within the Nordic/Baltic countries, children are treated according to the same protocol, i.e. NOPHO ALL-2008 protocol. Children and adolescents with Lymphoblastic Non-Hodgkin's Lymphoma (LBL) are treated in accordance with the EURO-LB 02 protocol, whereas adults with Lymphoblastic Non-Hodgkin's Lymphoma in Denmark are commonly treated in accordance with the NOPHO ALL-2008 protocol.

The longest treatment phase in both protocols is maintenance therapy, which is composed of 6-Mercaptopurine (6MP) and Methotrexate (MTX).

The cytotoxic property of 6MP relies upon conversion of 6MP into thioguanine nucleotides (TGN), which can be incorporated into DNA instead of guanine or adenine. This incorporation can cause nucleotide mismatching and cause cell death second to repetitive activation of the mismatch repair system. At Rigshospitalet investigators have developed pharmacological methods able to measure the incorporation of TGN into DNA (DNA-TGN). In a Nordic/Baltic study the investigators have demonstrated higher levels of DNA-TGN during maintenance therapy in children with ALL that do not develop relapse (Nielsen et al. Lancet Oncol. 2017 Apr;18(4)).

Preliminary studies indicate that the best approach to obtain DNA-TGN within a target range could be a combination of 6MP, MTX and 6-thioguanine (6TG), as 6TG more readily can be converted into TGN.

This study aims to explore if individual dose titration of 6TG added to 6MP/MTX therapy can achieve DNA-TGN levels above a set target above 500 fmol/µg DNA, and thus can be integrated into future ALL and LBL treatment strategies to reduce relapse rates in ALL and LBL.

The investigators plan to include 30 patients, and A) give incremental doses of 6TG until a mean DNA-TGN level above 500 fmol/µg DNA is obtained; and B) analyze the changes in DNA-TGN as well as cytosol levels of TGN and methylated 6MP metabolites (the latter inhibits purine de novo synthesis and thus enhance DNA-TGN incorporation), and C) occurrence of bone-marrow and liver toxicities during 6TG/6MP/MTX therapy.

DETAILED DESCRIPTION:
Acute Lymphoblastic Leukaemia (ALL) is the most frequent cancer in children. Each year approximately 220 children are diagnosed with ALL within the Nordic and Baltic countries.

The survival rate has improved significantly during the last decades, but the treatment still fails to cure approximately 15 % of the patients. A significant proportion of these relapses are likely to reflect adverse drug disposition rather than resistence to antileukemic agents. This emphazises the importance of developing new dosing strategies for reduction of relapse rates.

Most ALL relapses occur during or after maintenance therapy, and recent studies have indicated that almost 50% of these relapses are caused by insuffient exposure of DNA to the cytotoxic metabolites of 6MP.

Childhood Non-Hodgkin's Lymphoma (NHL) constitutes approximately 5% of all childhood malignancies in the Nordic countries and one out of four children with NHL has lymphoblastic lymphoma (LBL), the majority being T cell lymphoblastic lymphoma (T-LBL). Nordic children are treated in accordance with the EURO-LB 02 protocol, and every year 12-15 children are diagnosed with T-LBL within the Nordic countries. During the last 25 years, the cure rate for childhood T-LBL has increased from 25% to 75%, however, among patients failing first line therapy almost none survive.

The treatment of childhood and adolescent T-LBL and pre B cell lymphoblastic lymphoma (pB-LBL) resembles that of ALL and consists of an induction phase, a re-induction phase and a maintenance phase with oral 6MP/MTX, which is continued until 2 years from diagnosis to eliminate residual disease.

Adult LBL accounts for approximately 2% of all NHL, the majority being T-LBL (85-90%). LBL occurs more commonly in children than in adults, mostly in males, and has a highly aggressive nature. The prognosis in adults has dramatically improved with the introduction of pediatric intensive chemotherapy regimens for ALL, in concert with the prognosis of childhood NHL, with a disease-free survival reaching 45-72% in adults. However, a broadly accepted standard treatment for adult T- and pB-LBL has not yet been defined. Patients with T-LBL and pB-LBL, classified as non-HR, and in first remission will be eligible for inclusion into this study.

The cytotoxic property of 6MP relies upon conversion of 6MP into thioguanine nucleotides (TGN). TGN is a substrate for the DNA polymerase, and can be incorporated into DNA instead of guanosine or adenine (DNA-TGN). Incorporated TGN is hereafter occasionally mismatched to thymidine, which causes cell death second to activation of the mismatch repair system. During thiopurine-based therapy patients vary widely in their DNA-TGN levels and patients with low DNA-TGN levels may have an increased risk of relapse.

The investigators will explore

1. If individualized addition of 6TG to maintenance therapy can obtain a stable mean DNA-TGN level > 500 fmol/microgram DNA after addition of 6TG. DNA-TGN calculated as a 4 weeks mean.
2. The toxicities encountered during 6TG/6MP/MTX therapy.

The investigators hypothesize that 6TG/6MP/MTX combination therapy will achieve significantly higher DNA-TGN levels, and they will describe toxicities and thiopurine metabolite levels during MTX/6MP/6TG combination therapy.

The TEAM Study is designed as a prospective, multicentre, non-randomised, phase 1-2 clinical trial. This trial is a "proof of principle" and feasibility study planned with a modified crossover design, where participants serve as their own (historical) controls.

Additionally, data from the maintenance therapy substudy by Nielsen et. al (Lancet Oncol. 2017 Apr;18(4)) will be used in order to compare DNA-TG levels in patients receiving MTX/6MP based maintenance therapy, and DNA-TG levels in patients treated according to TEAM strategy (i.e. maintenance therapy with MTX/6MP/6TG).

Pharmacological target:

The investigators will include 30 participants. Upon inclusion in the TEAM study; 6MP dose is reduced to 2/3rd, if the current 6MP dose is > 50 mg/m2/day. However, if 6MP dose reduction is indicated, 6MP dose is not reduced below 50 mg/m2/day. If the current 6MP dose is < 50 mg/m2/day, the patient continues on this 6MP dose without dose reduction. 6TG treatment is initiated concomitantly. MTX dose is not changed. The investigators give A) incremental doses of 6TG (steps of 2.5 mg/meter square, max 12.5 mg/meter square) until a mean DNA-TGN of at least 500 fmol/µg DNA is obtained; and B) analyze the changes in DNA-TGN as well as Ery-TGN and MeMP. The dose increments of 6TG in steps of 2.5 mg/square metre will be spaced by intervals of at least two weeks, and DNA-TGN measurements will be measured weekly during 6TG dose increments. 6TG dose increments will continue until a mean DNA-TGN level > 500 fmol/µg or a maximum dose of 6TG of 12.5 mg/square metre is reached. If tolerated, the participant can then continue on that 6TG dose until the end of ALL/LBL therapy. Participants can at any time point drop out of TEAM by their own decision or by that of the treating physician. 6TG is provided as a liquid formulation to ease precise dose titration.

ELIGIBILITY:
Male and female patients of all ethnicities meeting all of the following criteria will be considered eligible for study participation:

1. Meet just one of the following:

   1. Confirmed diagnosis with non-HR-ALL and in first remission at inclusion into this investigation. Patients aged 1-45 years at diagnosis are eligible or
   2. Confirmed diagnosis with T-LBL or pB-LBL, and in first remission at inclusion into this investigation. Patients aged 0.6-45 years at the time of inclusion are eligible.
2. Have reached maintenance II therapy phase at inclusion.
3. Scheduled to receive 6MP/MTX maintenance therapy without any other concomitant myelosuppressive agents.
4. Patients must have a minimum of 3 months of 6MP/MTX maintenance therapy remaining at the time of inclusion.
5. Bilirubin < UNL according to age, factor 2-7-10 > 0.5 or INR < 1.5 within 1 week prior to inclusion.
6. WBC > 1.5 x109/L, ANC > 0.5 x109/L and TBC > 50 x109/L within 1 week prior to inclusion.
7. Subject, if female of child-bearing potential (defined as postmenarche), must present with a negative pregnancy test and must be nonlactating.
8. Sexually active females and males must use accepted safe contraception (OCPs, IUD, transdermal hormonal patch, vaginal hormonal ring or subdermal hormonal implants for women and condom for men) during therapy and until three months after study exit/early termination.
9. No live vaccines given within 2 months prior to inclusion.
10. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
11. Whenever appropriate, the child should participate in the oral and written informed consent process together with the parents. Involving the child in discussions and the decision-making process respects their emerging maturity. This process will be conducted with enough time and at the same time as obtaining the consent from the parents or the legal representative, so that the informed consent reflects the presumed will of the minor, in accordance with Article 4(a) of the Clinical Trial Directive.
12. If the study participant is unable to provide legally binding consent subject's legally authorized representative (e.g., both parent, legal guardian) must voluntarily sign and date a parental permission/ Informed Consent that is approved by the Danish Ethical Committee(EC), and the subject must sign an EC approved assent, before undergoing any protocol specific procedures or assessments according to Ethical considerations for clinical trials on medicinal products conducted with the paediatric population Directive 2001/20/EC1, ICH/GCP guidelines, and the Helsinki II Declaration.

Exclusion Criteria

1. Patients with ALL and a minimal residual disease (MRD)-negative bone-marrow at treatment day 29 (counted from diagnosis)-since these patients have an excellent prognosis on current therapy, and DNA-TG has not been associated with risk of relapse for these patients
2. 2. DNA-TG > 1,500 fmol/μg DNA due to (i) a potential association with toxicity (although not shown so far), and (ii) the lack of evidence regarding an association between reduced relapse rates and such high DNA-TG levels. If DNA-TG subsequently fell below 1,500 fmol/μg DNA, the patient would be eligible for TEAM.
3. Any clinical suspicion of relapse or disease progression on routine imaging or in laboratory results.
4. Previous sinusoidal obstruction syndrome (SOS) / veno-occlusive disease (VOD).
5. Allergic hypersensitivity towards any ingredients in the three medicinal products used in the study.

Ages: 6 Months to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Obtaining a stable mean DNA-TGN level > 500 fmol/microgram DNA after addition of 6TG. DNA-TGN calculated as a 4 weeks mean (maximum 6TG dose 12.5 mg/m.xq.). | From initiation of 6-thioguanine therapy until completion of ALL/LBL therapy
  After incremental doses in steps of 2.5 mg/m.sq. of 6-thioguanine at 2 weeks intervals up to a maximum dose of 12.5 mg/m.sq. or a dose-limiting toxicity occur or a mean DNA-TGN level above 500 fmol/microgram DNA is obtained. Maximum dose is expected to be reached within 10-12 weeks

SECONDARY OUTCOMES:
Erythrocyte 6MP cytosol metabolite levels | From initiation of 6-thioguanine therapy until completion of ALL/LBL therapy
  Erythrocyte levels are measured at 2 weeks intervals from initiation of 6-thioguanine therapy until completion of ALL/LBL therapy
Myelotoxicity | From initiation of 6-thioguanine therapy until completion of ALL/LBL therapy
  The dose-limiting toxicities are white blood cell count < 1.5x109/L and/or absolute neutrophil count < 0.5 x109/L and/or thrombocyte count < 50 x109/L),
Severe hepatotoxicity including sinusoidal obstruction syndrome | From initiation of 6-thioguanine therapy until completion of ALL/LBL therapy
  Dose-limiting severe hepatotoxicities include alanine aminotransferase > 20 x upper normal limit (UNL) and/or bilirubin > 3x UNL (according to age) and/or coagulation factors 2-7-10 < 0.50 (or INR > 1.5), and or clinical signs of sinusoidal obstruction syndrome (with at least 3 of 5 criteria: i) hepatomegaly, ii) hyperbilirubinaemia >UNL), iii) ascites, iv) weight gain of at least 5%, and v) thrombocytopenia (transfusion-resistant and/or otherwise unexplained by treatment induced myelosuppression.

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Schmiegelow, Professor, Study Chair — Department of Pediatrics and Adolescent Medicine. University Hospital Rigshospitalet, Copenhagen
Locations (4):
- Denmark (4):
  - Aarhus University Hospital Skejby, Skejby, Aarhus
  - Odense University Hospital, Dept. Pediatric Oncology, Odense, Odense C
  - Department of Pediatrics, Rigshospitalet, Copenhagen
  - Rigshospitalet, Department of Hematology, Copenhagen

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be entered into the Leukemia Registry of the Nordic Society of Pediatric Hematology/Oncology

REFERENCES:
- [Background] Gustafsson G, Schmiegelow K, Forestier E, Clausen N, Glomstein A, Jonmundsson G, Mellander L, Makipernaa A, Nygaard R, Saarinen-Pihkala UM. Improving outcome through two decades in childhood ALL in the Nordic countries: the impact of high-dose methotrexate in the reduction of CNS irradiation. Nordic Society of Pediatric Haematology and Oncology (NOPHO). Leukemia. 2000 Dec;14(12):2267-75. doi: 10.1038/sj.leu.2401961. PMID 11187918
- [Background] Schmiegelow K, Forestier E, Hellebostad M, Heyman M, Kristinsson J, Soderhall S, Taskinen M; Nordic Society of Paediatric Haematology and Oncology. Long-term results of NOPHO ALL-92 and ALL-2000 studies of childhood acute lymphoblastic leukemia. Leukemia. 2010 Feb;24(2):345-54. doi: 10.1038/leu.2009.251. Epub 2009 Dec 10. PMID 20010622
- [Background] Pui CH, Campana D, Evans WE. Childhood acute lymphoblastic leukaemia--current status and future perspectives. Lancet Oncol. 2001 Oct;2(10):597-607. doi: 10.1016/S1470-2045(01)00516-2. PMID 11902549
- [Background] Schmiegelow K, Nielsen SN, Frandsen TL, Nersting J. Mercaptopurine/Methotrexate maintenance therapy of childhood acute lymphoblastic leukemia: clinical facts and fiction. J Pediatr Hematol Oncol. 2014 Oct;36(7):503-17. doi: 10.1097/MPH.0000000000000206. PMID 24936744
- [Background] Relling MV, Hancock ML, Boyett JM, Pui CH, Evans WE. Prognostic importance of 6-mercaptopurine dose intensity in acute lymphoblastic leukemia. Blood. 1999 May 1;93(9):2817-23. PMID 10216075
- [Background] Schmiegelow K, Schroder H, Gustafsson G, Kristinsson J, Glomstein A, Salmi T, Wranne L. Risk of relapse in childhood acute lymphoblastic leukemia is related to RBC methotrexate and mercaptopurine metabolites during maintenance chemotherapy. Nordic Society for Pediatric Hematology and Oncology. J Clin Oncol. 1995 Feb;13(2):345-51. doi: 10.1200/JCO.1995.13.2.345. PMID 7531219
- [Background] Schmiegelow K, Forestier E, Kristinsson J, Soderhall S, Vettenranta K, Weinshilboum R, Wesenberg F; Nordic Society of Paediatric Haematology and Oncology. Thiopurine methyltransferase activity is related to the risk of relapse of childhood acute lymphoblastic leukemia: results from the NOPHO ALL-92 study. Leukemia. 2009 Mar;23(3):557-64. doi: 10.1038/leu.2008.316. Epub 2008 Nov 6. PMID 18987654
- [Background] Cooper SL, Brown PA. Treatment of pediatric acute lymphoblastic leukemia. Pediatr Clin North Am. 2015 Feb;62(1):61-73. doi: 10.1016/j.pcl.2014.09.006. Epub 2014 Oct 18. PMID 25435112
- [Background] Hunger SP, Winick NJ, Sather HN, Carroll WL. Therapy of low-risk subsets of childhood acute lymphoblastic leukemia: when do we say enough? Pediatr Blood Cancer. 2005 Dec;45(7):876-80. doi: 10.1002/pbc.20501. No abstract available. PMID 16007585
- [Background] Karran P, Attard N. Thiopurines in current medical practice: molecular mechanisms and contributions to therapy-related cancer. Nat Rev Cancer. 2008 Jan;8(1):24-36. doi: 10.1038/nrc2292. PMID 18097462
- [Background] Hedeland RL, Hvidt K, Nersting J, Rosthoj S, Dalhoff K, Lausen B, Schmiegelow K. DNA incorporation of 6-thioguanine nucleotides during maintenance therapy of childhood acute lymphoblastic leukaemia and non-Hodgkin lymphoma. Cancer Chemother Pharmacol. 2010 Aug;66(3):485-91. doi: 10.1007/s00280-009-1184-5. Epub 2009 Dec 3. PMID 19956952
- [Background] Ebbesen MS, Nersting J, Jacobsen JH, Frandsen TL, Vettenranta K, Abramsson J, Wesenberg F, Schmiegelow K. Incorporation of 6-thioguanine nucleotides into DNA during maintenance therapy of childhood acute lymphoblastic leukemia-the influence of thiopurine methyltransferase genotypes. J Clin Pharmacol. 2013 Jun;53(6):670-4. doi: 10.1002/jcph.81. Epub 2013 Apr 15. No abstract available. PMID 23585236
- [Background] Jacobsen JH, Schmiegelow K, Nersting J. Liquid chromatography-tandem mass spectrometry quantification of 6-thioguanine in DNA using endogenous guanine as internal standard. J Chromatogr B Analyt Technol Biomed Life Sci. 2012 Jan 15;881-882:115-8. doi: 10.1016/j.jchromb.2011.11.032. Epub 2011 Nov 28. PMID 22178190
- [Background] Erb N, Harms DO, Janka-Schaub G. Pharmacokinetics and metabolism of thiopurines in children with acute lymphoblastic leukemia receiving 6-thioguanine versus 6-mercaptopurine. Cancer Chemother Pharmacol. 1998;42(4):266-72. doi: 10.1007/s002800050816. PMID 9744770
- [Background] Schmiegelow K, Bjork O, Glomstein A, Gustafsson G, Keiding N, Kristinsson J, Makipernaa A, Rosthoj S, Szumlanski C, Sorensen TM, Weinshilboum R. Intensification of mercaptopurine/methotrexate maintenance chemotherapy may increase the risk of relapse for some children with acute lymphoblastic leukemia. J Clin Oncol. 2003 Apr 1;21(7):1332-9. doi: 10.1200/JCO.2003.04.039. PMID 12663723
- [Background] Nygaard U, Toft N, Schmiegelow K. Methylated metabolites of 6-mercaptopurine are associated with hepatotoxicity. Clin Pharmacol Ther. 2004 Apr;75(4):274-81. doi: 10.1016/j.clpt.2003.12.001. PMID 15060506
- [Background] Nielsen SN, Frandsen TL, Nersting J, Hjalgrim LL, Schmiegelow K. Pharmacokinetics of 6-Thioguanine and 6-Mercaptopurine Combination Maintenance Therapy of Childhood ALL: Hypothesis and Case Report. J Pediatr Hematol Oncol. 2015 Apr;37(3):e206-9. doi: 10.1097/MPH.0000000000000246. PMID 25171455
- [Background] Escherich G, Richards S, Stork LC, Vora AJ; Childhood Acute Lymphoblastic Leukaemia Collaborative Group (CALLCG). Meta-analysis of randomised trials comparing thiopurines in childhood acute lymphoblastic leukaemia. Leukemia. 2011 Jun;25(6):953-9. doi: 10.1038/leu.2011.37. Epub 2011 Mar 4. PMID 21372841
- [Background] Stork LC, Matloub Y, Broxson E, La M, Yanofsky R, Sather H, Hutchinson R, Heerema NA, Sorrell AD, Masterson M, Bleyer A, Gaynon PS. Oral 6-mercaptopurine versus oral 6-thioguanine and veno-occlusive disease in children with standard-risk acute lymphoblastic leukemia: report of the Children's Oncology Group CCG-1952 clinical trial. Blood. 2010 Apr 8;115(14):2740-8. doi: 10.1182/blood-2009-07-230656. Epub 2010 Feb 1. PMID 20124218
- [Background] Lancaster DL, Lennard L, Rowland K, Vora AJ, Lilleyman JS. Thioguanine versus mercaptopurine for therapy of childhood lymphoblastic leukaemia: a comparison of haematological toxicity and drug metabolite concentrations. Br J Haematol. 1998 Jul;102(2):439-43. doi: 10.1046/j.1365-2141.1998.00812.x. PMID 9695957
- [Background] Nielsen SN, Grell K, Nersting J, Frandsen TL, Hjalgrim LL, Schmiegelow K. Measures of 6-mercaptopurine and methotrexate maintenance therapy intensity in childhood acute lymphoblastic leukemia. Cancer Chemother Pharmacol. 2016 Nov;78(5):983-994. doi: 10.1007/s00280-016-3151-2. Epub 2016 Sep 6. PMID 27600880
- [Background] Nielsen SN, Grell K, Nersting J, Abrahamsson J, Lund B, Kanerva J, Jonsson OG, Vaitkeviciene G, Pruunsild K, Hjalgrim LL, Schmiegelow K. DNA-thioguanine nucleotide concentration and relapse-free survival during maintenance therapy of childhood acute lymphoblastic leukaemia (NOPHO ALL2008): a prospective substudy of a phase 3 trial. Lancet Oncol. 2017 Apr;18(4):515-524. doi: 10.1016/S1470-2045(17)30154-7. Epub 2017 Mar 1. PMID 28258828